CLINICAL TRIAL: NCT07289217
Title: A Randomized Controlled Decentralized Clinical Pilot Trial to Assess the Effectiveness and Sagety of the Digital Cognitive Behavioral Therapy Intervention SleepQ for Insomnia
Brief Title: WELT-REST: WELT Randomized Evaluation of Sleep Therapy
Acronym: WELT-REST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WELT corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCTP-DI-A-01
Record Dates: First submitted 2025-12-03; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: dCBT - I; CBT - I; Insomnia; Cognitive Behavioral Therapy; Sleep Disorder; Digital Therapeutics; Digital CBT - I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SleepQ Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) (Experimental)
  Interventions: Behavioral: SleepQ Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I)
- Care-as-Usual (CAU) (No Intervention)

INTERVENTIONS:
Behavioral: SleepQ Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) — SleepQ is a fully digital, individualized 12-week cognitive behavioral therapy program for adults with insomnia. The intervention is delivered via the SleepQ mobile application and includes structured CBT-I components such as sleep restriction therapy, stimulus control, psychoeducation, cognitive restructuring, sleep hygiene training, and daily sleep diary input, in addition to Care-as-Usual (CAU).
  Arms: SleepQ Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I)

SUMMARY:
The goal of this clinical trial is to learn whether the SleepQ mobile app can help reduce insomnia symptoms in adults diagnosed with insomnia. The main questions it aims to answer are:

* Does adding the SleepQ app to care as usual (CAU) improve insomnia symptoms after 12 weeks?
* Does SleepQ also improve depressive symptoms, anxiety, beliefs about sleep and daily functioning?

Researchers will compare CAU + SleepQ to CAU alone to see whether SleepQ provides additional benefits for sleep and well-being.

Participants will take part remotely from home, be randomly assigned to either SleepQ+CAU or CAU alone, and complete online questionnaires at baseline, week 6, and week 12 about their sleep, mood, and daily functioning.

Participants in the intervention group will use the SleepQ app for 12 weeks while continuing their usual care.

DETAILED DESCRIPTION:
SleepQ is digital CBT-I application developed to align with national clinical guidelines for the treatment of sleep disorders. The program includes psychoeducation, sleep restriction therapy, stimulus control, sleep hygiene approaches, cognitive restructuring, and relaxation exercises. The app also incorporates a digital sleep diary, personalized sleep timing recommendations, interactive learning modules, quizzes to reinforce concepts, and monitoring of therapy progress. The overall design aims to support engagement and autonomous adherence to CBT-I principles by providing step-by-step guidance and feedback throughout the therapeutic course.

The pilot clinical trial will evaluate the effectiveness of SleepQ as an add-on to care as usual (CAU) compared with CAU alone in adults diagnosed with insomnia. Approximately 80 adult participants with a confirmed diagnosis of insomnia will be enrolled and randomized in a 1:1 ratio to the intervention group (SleepQ + CAU) or the control group (CAU alone). The study will be conducted as a fully decentralized trial within Germany. Screening, informed consent, eligibility confirmation, randomization, and all outcome assessments will be conducted remotely. Participants will complete self-reported questionnaires at baseline, week 6, and week 12 to assess changes in insomnia severity and related symptoms.

The primary endpoint is the reduction in insomnia symptoms after 12 weeks, and secondary outcomes include changes in depressiv symptoms, anxiety, dysfunctional beliefs about sleep, and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old
* Confirmed current diagnosis of F51.0 Nonorganic insomnia or G47.0 Sleep disorders
* Possession of a mobile device with internet connection (must be run on iOS software, minimum version 18) with internet connection
* Sufficient German language proficiency required for the correct use of the intervention and the mobile device
* Personal e-mail address for registration
* Willing and able to provide written informed consent
* Insomnia Severity Index (ISI) socre of 15 or higher, indicating clinically relevant symptoms of insomnia
* Registered with a GP, sleep specialist or other health care professional

Exclusion Criteria:

* Use of a digital interventioan for insomnia treatment in the past 6 months or planned use of comparable digital intervention during the study period
* PHQ-9 score at screening ≥ 20 and/or item 9 f PHQ-9 ≥ 1
* GAD-7 score at screening ≥ 15
* Intermittent use and/or recent initiation (< 3m) or planned use of insomnia specific prescription-only pharmacological therapy
* Intermittent use and/or recent initiation (< 3m) or planned use of a psychotropic during the study period which has recognised potential effects on insomnia
* Participation in CBT or other psychotherapy to treat sleep disorders in the last 6 months (outpatient, inpatient) or planned start during the study period
* Known history or diagnosis of substance or alchol abuse or dependence within 12 months prior to screening (diagnosis of F10-F19, excluding F17.1 and F17.2)
* Current or planned participation in other clinical trials during the study period
* Working in shifts
* Currently pregnant or planning to become pregnant within the next 3 months
* Any surgical procedure that was scheduled, planned, or conducted within the timeframe of the study (minor outpatient procedures under local anaesthetic or with no anesthetic are permitted)
* Diagnosis of epilepsy
* Presence of serious mental illness, such as (schizophrenia F 20.-, acute transient psychotic disorders F23.-, active manic episode F30.-, bipolar disorder F31.-, severe depression F32.3, F33.3)
* Other diseases (such as acute or severe cardiac diseases, acute or severe respiratory diseases, acute or severe gastrointestinal diseases), conditions or therapies which, in the opinion of the investigator, could confound the study results or contraindicate participation.
* Acute suicidal thoughts or intentions within the past 12 months
* Presence of obstructive sleep apnea, restless legs syndrome, parasomnia, and other sleep behavior problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Score from Baseline to Week 12 | From baseline to 12 weeks after enrollment
  The Insomnia Severity Index (ISI) is a 7-item validated self-report questionnaire assessing the severity and impact of insomnia symptoms. Total scores range from 0 to 28, with higher scores indicating more severe insomnia. ISI is administered at baseline and week 12. The outcom is calculated a the change in total ISI score from baseline to week 12.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) Score from Baseline to Week 12 | From baseline to week 12
  The PHQ-9 is a 9-item validated self-report measure of depressive symptoms. Each item is scored from 0 to 3, producing a total score from 0 to 27, with higher scores indicating more severe depression. The outcome is the change in total PHQ-9 score from baseline to week 12.
Change in Generalized Anxiety Disorder-7 (GAD-7) Score from Baseline to Week 12 | From baseline to week 12
  The GAD-7 is a 7-item validated self-report measure of anxiety symptoms. Each item is scored from 0 to 3, yielding a total score from 0 to 21, with higher scores indicating more severe anxiety. The outcome is the change in total GAD-7 score from baseline to week 12.
Change in Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) Score from Baseline to Week 12 | From baseline to week 12
  The DBAS-16 is a 16-item self-report scale assessing maladaptive sleep-related beliefs. Items are rated from 0 (strongly disagree) to 10 (strongly agree). The total score is the mean of all items and ranges from 0 to 10, with higher scores indicating stronger dysfunctional beliefs. The outcome is the change in mean DBAS-16 score from baseline to week 12.
Change in Work and Social Adjustment Scale (WSAS) Score from Baseline to Week 12 | From baseline to week 12
  The WSAS is a 5-item self-report measure assessing functional impairment across work, home management, social activities, and relationships. Each item is scored from 0 (no impairment) to 8 (severe impairment), producing a total score from 0 to 40. Higher scores indicate greater functional impairment. The outcome is the change in total WSAS score from baseline to week 12.
Change in EuroQol Visual Analog Scale (EQ-VAS) Score from Baseline to Week 12 | From baseline to week 12
  The EQ-VAS is a self-rated measure of overall health-related quality of life. Participants rate their current health on a 0 to 100 visual analog scale, where 0 indicates the worst imaginable health and 100 the best imaginable health. The outcome is the change in EQ-VAS score from baseline to week 12.

OTHER OUTCOMES:
Change in Patient Satisfaction With the SleepQ App From Intervention Start to Week 12 | From intervention start (code activation) to week 12
  Patient satisfaction with the SleepQ digital intervention will be assessed in the intervention group using a validated satisfaction quesitonnaire based on the Second Ordinance Amending the Digital Health Applications Ordinance (BfArM, 2025)
  The questionnaire includes five items rated on a 0-10 Likert-type scale:
  1. I was able to easily understand the DiGA.
  2. The DiGA functioned reliably.
  3. When I had questions, I received support easily and without complications.
  4. The DiGA helped me understand my condition better than before.
  5. How likely is it that you would recommend this DiGA to friends and family?
  For Items 1-4, higher scores indicate stronger agreement (0 = does not apply at all; 10 = extremely likely).
  For Item 5, higher scores indicate greater likelihood of recommendation (0 = extremely unlikely; 10 = extremely likely).
  Scores will be analyzed as change from intervention start.

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin Medical Association (Ärztekammer Berlin), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided